CLINICAL TRIAL: NCT04592484
Title: A First-in-Human Study of CDK-002 (exoSTING) in Subjects With Advanced/Metastatic, Recurrent, Injectable Solid Tumors, With Emphasis on Squamous Cell Carcinoma of the Head and Neck, Triple Negative Breast Cancer, Anaplastic Thyroid Carcinoma, and Cutaneous Squamous Cell Carcinoma
Brief Title: A First-in-Human Study of CDK-002 (exoSTING) in Subjects With Advanced/Metastatic, Recurrent, Injectable Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Codiak BioSciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDK-002-101
Record Dates: First submitted 2020-08-18; First posted 2020-10-19 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CDK-002 (Experimental)
  Interventions: Biological: CDK-002

INTERVENTIONS:
Biological: CDK-002 — CDK-002 administered intratumorally

SUMMARY:
This is a first-in-human, Phase 1/2 open-label, multicenter, dose escalation, safety, pharmacodynamic, and PK study of CDK-002 in subjects with advanced/metastatic, recurrent, injectable solid tumors, whose disease has progressed despite receiving standard of care treatment. CDK 002 will be administered intratumorally (IT).

Part A will enroll subjects with advanced/metastatic, recurrent, injectable solid tumors with emphasis on head and neck squamous cell cancer (HNSCC), triple negative breast cancer (TNBC), anaplastic thyroid carcinoma (ATC) and cutaneous squamous cell carcinoma (cSCC).

ELIGIBILITY:
Inclusion Criteria:

Criteria for Inclusion:

1. Age ≥ 18 years at the time of signing the informed consent form.
2. Histologically confirmed advanced, recurrent or metastatic injectable solid tumor and has received the following prior therapy:

   1. HNSCC: Subject must have been previously treated with a platinum-based chemotherapy regimen and/or a programmed cell death-protein 1 (PD-1) inhibitor.
   2. TNBC: Subject must have been treated with at least 1 chemotherapy regimen and/or PD-L1 or PD-1 inhibitor for metastatic disease.
   3. ATC: Subject must be considered inoperable and not considered to benefit from additional chemotherapy and/or radiation.
   4. cSCC: Subject must have previously been treated with radiation therapy and/or chemotherapy and/or PD-L1 or PD-1 inhibitor.
   5. Subjects with other advanced solid tumors that have progressed following standard therapy or for which there is no standard of care therapy with an overall survival (OS) benefit.
3. Measurable disease per RECIST v1.1 and ≥1 lesion that is measurable (ie, ≥1.0 cm by CT, MRI, or ruler or caliper measurements for cutaneous lesions or other superficial lesions in longest diameter [non-lymph nodes] or ≥1.5 cm in shortest diameter for lymph nodes) and amenable to tumoral injection and biopsy per Investigator assessment.
4. Agrees to have a pre-treatment tumor biopsy within 7 days prior to the first dose of CDK-002, and 2 on-treatment tumor biopsies of the same lesion. Biopsies may be core needle, incisional, or excisional biopsies. For cutaneous lesions, a punch biopsy may be acceptable. Fine needle aspiration (FNA) is not acceptable.
5. Understands and can comply with the study requirements and has signed the informed consent form.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
7. Life expectancy of at least 3 months.
8. Acceptable liver function.
9. Acceptable renal function.
10. Acceptable hematologic status.
11. Negative serum pregnancy test (for women of child-bearing potential) within 72 hours before the first dose of CDK-002.

Exclusion Criteria:

Criteria for Exclusion:

1. Prior treatment with a STING agonist.
2. Cytotoxic chemotherapy, biologic agents, investigational agents, or radiation therapy within 4 weeks prior to the first dose of CDK 002 (6 weeks for nitrosoureas or mitomycin C). The interval can be reduced to 2 weeks for bone-only radiation therapy.
3. Small-molecule kinase inhibitors or hormonal anticancer agents within 14 days prior to the first dose of CDK 002.
4. Clinically significant ongoing AEs that have not returned to baseline or to Grade 1 NCI CTCAE v5.0.
5. Immunosuppressive agents including corticosteroids within 14 days of first dose of CDK 002. Topical, intranasal or inhaled corticosteroids, physiologic doses of systemic steroids or limited treatment with systemic steroids (ie, for IV contrast prophylaxis) may be administered with Sponsor approval.
6. Major surgery within 6 weeks or minor surgery (excluding tumor biopsies) within 14 days prior to the first dose of CDK 002 or if subject has not clinically recovered.
7. Clinically active central nervous system (CNS) metastases or carcinomatous meningitis. Subjects with stable brain metastasis may be enrolled with Sponsor approval.
8. Metastatic liver involvement that exceeds one-third of total liver volume.
9. Clinically significant cardiovascular disease including but not limited to New York Heart Association Class III or IV heart failure, myocardial infarction or stroke within the past 6 months prior to the first dose of CDK 002, uncontrolled arrhythmia, or severe aortic stenosis. Sponsor approval of subjects with an arrhythmia is required.
10. History of myocarditis.
11. Active, uncontrolled bacterial, viral, or fungal infections requiring systemic therapy. Prophylactic antibiotics are acceptable.
12. Prior organ or stem cell transplant.
13. Primary immune deficiency.
14. Pregnant or nursing women.
15. Active Hepatitis B or C infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of ascending doses of CDK-002 | up to 2 years
  Incidence of treatment-emergent adverse events as assessed by CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Roger Cohen, MD, Principal Investigator — University of Pennsylvania Hospital
Locations (8):
- United States (4):
  - Honor Health, Scottsdale, Arizona
  - Columbia University/CUMC, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - NEXT Oncology, San Antonio, Texas
- United Kingdom (4):
  - The Beatson West of Scotland Cancer Centre/ Gartnavel General Hospital, Glasgow
  - Oxford University Hospitals NHS Trust, Headington
  - The Royal Marsden Hospital, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No